CLINICAL TRIAL: NCT04875624
Title: Neurodevelopmental Outcome of Normoglycemic Versus Hypoglycemic Neonates at Risk for Hypoglycemia
Brief Title: Neurodevelopment of Hypoglycemic Neonates
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-13030
Record Dates: First submitted 2021-04-29; First posted 2021-05-06 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Neonatal Hypoglycemia; Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypoglycemic neonates: Preterm or small for gestational age neonates at risk for hypoglycemia who were found to be hypoglycemic during the screening for hypoglycemia
  Interventions: Diagnostic Test: Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-4)
- Normoglycemic neonates: Preterm or small for gestational age neonates who were found to be normoglycemic during the screening for hypoglycemia
  Interventions: Diagnostic Test: Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-4)

INTERVENTIONS:
Diagnostic Test: Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-4) — Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-4) will be administered by one of the 2 blinded examiners who are unaware of neonatal glycemia status. Bayley-4 examines Cognitive, Language, Motor, Social-Emotional and Adaptive Behavior domains of development and may require up to 120 minutes to complete.

SUMMARY:
The investigators propose to prospectively conduct a neurodevelopmental evaluation of SGA and late preterm neonates who underwent risk-based screening for hypoglycemia at newborn nursery during the first 24 hours of life based on AAP (American Academy of Pediatrics) hypoglycemia guidelines at 18 to 24 months of age. As per internal neonatal unit protocol (reflecting AAP guidelines), all neonates at risk of hypoglycemia (all preterm infants, term infants who are SGA or LGA and IDM) are routinely screened for hypoglycemia during the first 24 hours of life via bedside point of care glucose devices (see attached Weiler neonatal intensive care unit (NICU) hypoglycemia screening protocol). The investigators will compare neurodevelopmental outcomes of those who were and were not hypoglycemic in the newborn nursery based on electronic health record data.

DETAILED DESCRIPTION:
Neonatal hypoglycemia is the most common metabolic problem in neonates and a preventable cause of brain injury in infancy. Key risk factors for neonatal hypoglycemia include being born preterm, small for gestational age (SGA), large for gestational age (LGA), and being an infant of a diabetic mother (IDM) (1). Approximately 30% of all neonates are considered at risk, of whom approximately 50% develop hypoglycemia (2). Neonatal hypoglycemia is tightly related to adverse neurodevelopmental and brain injury outcomes, particularly among preterm infants who are SGA (3). Screening is recommended for babies with known risk factors (4). Glucose is an essential molecule that supplies energy for brain consumption. Neurons and glial cells in the brain are sensitive to hypoglycemia. Neonatal hypoglycemia has been recognized as a cause of long-term severe neurologic and neurodevelopmental morbidity due to damage to these cells (5). Neonatal hypoglycemia is a common finding associated with brain injury, neurodevelopmental delay, visual impairment, and behavioral problems.

Management of hypoglycemia in the newborn period is highly variable among institutions, and recommendations from different professional societies vary. In 2011, the American Academy of Pediatrics (AAP) Committee on Fetus and Newborn published a clinical report suggesting management guidelines for late-preterm and term infants with associated risk factors, targeting infants of IDM, LGA and SGA neonates (2). Of note, AAP clinical report provides guidelines only for the initial 24 hours of life and recommends screening of IDM and LGA infants for 12 hours and screening of SGA and late preterm infants for 24 hours. Canadian Paediatric Society in their updated position statement recommends a similar screening algorithm based on risk factors, stressing the importance of adequate feeding in SGA and late preterm infants. The Pediatric Endocrine Society (PES) issued the recommendations for evaluation and management of persistent hypoglycemia in neonates, infants and children beyond the initial 24 hours of life. The 2011 AAP guidelines define neonatal hypoglycemia as blood glucose <47 mg/dL and recommend maintaining blood glucose >40 mg/dL in the first 4 hours and >45 mg/dl between hours 4-24 (6). The PES has an even stricter threshold of >50 mg/dL. The AAP guidance, however, applies only to the first 24 hours of life, and the PES strategy focuses on infants beyond 48 hours of life with persistent hypoglycemia (7).

Due to poor correlation between blood glucose concentrations, clinical manifestations and controversial treatment thresholds, it is difficult to define a safe blood glucose level. Several studies have analyzed the effects of various ranges of hypoglycemia on neurodevelopmental outcome. However, variable results regarding the effect of hypoglycemia on the neurodevelopmental outcome have been reported without any clear conclusion (5,8-12).

In this study investigators propose to prospectively conduct a neurodevelopmental evaluation of SGA and late preterm neonates who underwent risk-based screening for hypoglycemia at newborn nursery during the first 24 hours of life based on AAP hypoglycemia guidelines at 18 to 24 months of age. As per neonatal unit protocol (reflecting AAP guidelines), all neonates at risk of hypoglycemia (all preterm infants, term infants who are SGA or LGA and IDM) are routinely screened for hypoglycemia during the first 24 hours of life via bedside point of care glucose devices (see attached Weiler NICU hypoglycemia screening protocol).

Aims:

1. To compare cognitive and motor development assessed with the Bayley-4 scoring system between the normoglycemic and hypoglycemic at-risk SGA/late preterm neonates
2. To assess language development, social-emotional and adaptive behavior in the normoglycemic and hypoglycemic at-risk neonates
3. To compare Bayley-4 scores between the cohort of neonates needing intravenous (IV) dextrose administration/neonatal intensive care admission to those with hypoglycemia managed in the newborn nursery as well as to those neonates who remained normoglycemic

Hypothesis:

The investigators hypothesize that SGA and late preterm hypoglycemic neonates admitted to newborn nursery will have inferior neurodevelopmental outcome at 18 to 24 months age when compared to SGA and late preterm infants with normoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Born at 35 weeks or more of gestation
* Birth weight of 2000 g or more
* Indication for routine screening for hypoglycemia: late preterm infants (gestational age from 35 weeks 0 days to 36 weeks 6 days) and newborns who were SGA (birth weight below the 10th percentile on the 2013 Fenton curve).

Exclusion Criteria:

* Neonates with indication for hypoglycemia screening - screening not properly done or missing
* Unable to reach the subject for neurodevelopmental assessment
* Non-English speaking subjects

Ages: 18 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a cross-sectional study evaluating neurodevelopmental outcome at 18 to 24 months of SGA/late preterm neonates who received risk-based screening for hypoglycemia and were found to be either normoglycemic or hypoglycemic during hospitalization. Eligible subjects will be identified via electronic health record search, and their hypoglycemia risk factors will be verified together with glycemia status. Parents of eligible subjects will be contacted via phone and invited for research participation; Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-4) will be administered by one of the 2 blinded examiners who are unaware of neonatal glycemia status. Bayley-4 examines Cognitive, Language, Motor, Social-Emotional and Adaptive Behavior domains of development .
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Comparison of cognitive development using Bayley-4 scoring system | 120 minutes
  Compare cognitive development assessed with the Bayley-4 scoring system between the normoglycemic and hypoglycemic at-risk SGA/late preterm neonates
Comparison of motor development using Bayley-4 scoring system | 120 minutes
  Assess motor development between the normoglycemic and hypoglycemic at-risk neonates

SECONDARY OUTCOMES:
Comparison of language development using Bayley-4 scoring system | 120 minutes
  Compare language development using Bayley-4 scoring system between the normoglycemic and hypoglycemic at-risk neonates
Comparison of social-emotional behavior using Bayley-4 scoring system | 120 minutes
  Comparison of social-emotional behavior using Bayley-4 scoring system between the normoglycemic and hypoglycemic at-risk neonates
Comparison of adaptive behavior using Bayley-4 scoring system | 120 minutes
  Comparison of adaptive behavior using Bayley-4 scoring system between the normoglycemic and hypoglycemic at-risk neonates

CONTACTS AND LOCATIONS:
Overall Officials: Jillian Connors, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, Weiler Hospital, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No